CLINICAL TRIAL: NCT06111222
Title: Multicentric Prospective Study on the Visual Performance of Patients Implanted With a Multifocal Intraocular Lens
Brief Title: Visual Performance of Patients Implanted With a Multifocal IOL
Acronym: VISUAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPAS-SUR-021-01
Record Dates: First submitted 2023-10-18; First posted 2023-11-01 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cataract; Refractive Lens Exchange
Keywords: cataract; multifocal IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Patients scheduled for cataract or refractive lens exchange surgery requiring bilateral implantation of multifocal IOL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bilateral implantation of investigational device (Other): Bilateral implantation of investigational device
  Interventions: Device: AT ELANA

INTERVENTIONS:
Device: AT ELANA — The device is CE-approved. The device is a posterior chamber multifocal intraocular lens (IOL) indicated for aphakia after surgical extraction of the cataractous natural lens. The device is also indicated for non-cataractous, presbyopic patients (PRELEX) who seek greater independence from glasses for intermediate and/or near distances. It is an aspheric (aberration-neutral) IOL made of hydrophobic acrylic material, coated with heparin with modified C-loop haptics.

SUMMARY:
The goal of this clinical trial is to learn about the visual performance of a new multifocal intra-ocular lens in patients presenting for cataract or refractive lens exchange surgery. The main question it aims to answer is: What is the visual performance and patient satisfaction twelve months post-operatively? Participants will receive bilateral implantation of the investigational device, undergo post-operative assessments, and provide feedback on their overall visual satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Patients scheduled for bilateral AT ELANA 841P phacoemulsification cataract extraction or Femtosecond-Laser-Assisted-Cataract-Surgery (cataract grades of 1, 2, 3 on the LOCSIII scale) and IOL implantation (Cataract or PRELEX) with a maximum of 28 days between both implantations; Calculated IOL power within the limited IOL Diopter range of +15.0D to +27.0D
* No visual acuity limiting pathologies other than cataract;
* Corneal Astigmatism of <1.0 D;
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures;
* Written informed consent for participation in the study and data protection.

Exclusion Criteria:

* Corneal Astigmatism of ≥1.0 D;
* Difficulty for cooperation (distance from their home, general health conditions);
* History of acute or chronic disease, pathology, illness, or ocular trauma that would, in the surgeon's opinion, confound results (e.g., corneal pathology, OHT, glaucoma suspect, glaucoma, macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, amblyopia, etc.);
* Visual field loss which has an impact on visual acuity;
* Use of systemic or ocular medication that might affect vision;
* Patients with amblyopia, strabismus, forme fruste keratoconus or keratoconus;
* Pupil abnormalities (non-reactive, tonic pupils, abnormal myosis or mydriasis, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions);
* Capsular or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g., pseudoexfoliation syndrome);
* Cataract grades of 4, 5 or 6 on the LOCSIII scale ;
* Surgeries with incision size of ≥2.75mm ;
* Immediate Sequential Bilateral Cataract Surgery ;
* Concurrent participation in another device investigation;
* Usage of contact lenses during participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mean monocular best-corrected distance visual acuity (CDVA) | Three (3) Months
  The objective is to evaluate Corrected Distance Visual Acuity (CDVA)

SECONDARY OUTCOMES:
Refractive Predictability / Manifest Refraction and Prediction Error | Twelve (12) Months
  Descriptive analysis of the manifest refraction parameters sphere, cylinder, and spherical equivalent (MRSE) will be reported to determine refractive predictability

OTHER OUTCOMES:
Uncorrected Visual Acuities | Twelve (12) Months
  Binocular uncorrected distance, intermediate and near visual acuity (UDVA, UIVA, UNVA)
Corrected Distance Visual Acuities | Twelve (12) Months
  Best-corrected monocular and binocular distance visual acuity (CDVA)
Corrected Intermediate and Near Visual Acuities | Twelve (12) Months
  Binocular Distance-corrected intermediate and near visual acuity
Refractive predictability | Twelve (12) Months
Patient Reported Outcome Measures (PROMs) | Three (3) Months
Postoperative use of spectacles | Twelve (12) Months
Defocus Curves | Twelve (12) Months
  Monocular and Binocular
Binocular Contrast Sensitivity | Twelve (12) Months
  Photopic and Mesopic
Posterior Capsule Opacification (PCO) | Twelve (12) Months
Nd:YAG rate | Twelve (12) Months
  Incidence of Neodymium:yttrium-aluminum-garnet (Nd:YAG) laser capsulotomy as treatment for PCO
Optimization of CZM IOL calculation tools | Twelve (12) Months
  Anonymized Biometry raw data will be collected and used to optimize Carl ZEISS Meditec IOL calculation tools, such as the ZEISS IOL Power Calculation Service and algorithms of the optical biometer IOL Master 700, to improve future clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (2):
  - Universitätsklinikum Heidelberg, Heidelberg
  - PVK Precise Vision GmbH, Rheine
- Ofatlivist Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No